CLINICAL TRIAL: NCT05379946
Title: A Phase 1/2, Open Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of D-1553 in Combination With IN10018 in Subjects With Advanced or Metastatic Solid Tumors With KRasG12C Mutation
Brief Title: Study to Evaluate D-1553 in Combination With IN10018 in Subjects With Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Collaborators: InxMed (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D1553-106
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1b Dose escalation of D-1553 plus IN10018 (Experimental): Phase 1b will evaluate up sequential cohorts with different doses of IN10018 together with D-1553 to determine safety, tolerability, MTD and RDE in patients with solid tumors with KRasG12C mutation.
  Interventions: Drug: D-1553; Drug: IN10018
- Phase 2 Doseexpansion of D-1553 plus IN10018 (Experimental): Phase 2 will include more subjects to further evaluate the safety and efficacy of D-1553 in combination with IN10018 in patients with solid tumors with KRasG12C mutation.
  Interventions: Drug: D-1553; Drug: IN10018

INTERVENTIONS:
Drug: D-1553 — D-1553 is a oral dosed novel, targeted KRasG12C inhibitor that is being developed as a potential oral agent for advanced or metastatic solid tumors with KRasG12C mutation
Drug: IN10018 — IN10018 orally once daily at approximately the same time each day

SUMMARY:
This is a phase 1/2, open label study of D-1553 in combination with IN10018 to assess the safety and tolerability, identify the MTD and RP2D, evaluate the PK properties and antitumor activities in subjects with advanced or metastatic solid tumor with KRasG12C mutation

ELIGIBILITY:
Inclusion Criteria:

* Subject with histologically proven, locally advanced, unresectable and/or metastatic solid tumor, for which no standard treatment is available or the subject is refractory to or intolerant of existing standard treatment.
* Subject has KRasG12C mutation in tumor tissue or other biospecimens (only for phase1b) containing cancer cells or DNA. Historical, local laboratory result (up to 5 years prior to this study) can be used.
* Subject has tumor type requirement as follows: advanced or metastatic solid tumors including NSCLC and CRC.
* Subject has measurable disease according to RECIST, v1.1

Exclusion Criteria:

Subject with unstable or progressive central nervous system (CNS) metastases.

* Subject with acute myocardial infarction, severe/unstable angina; or with cardiac insufficiency of New York Heart Association Functional Classification Grade 2 or above.
* Subject has corrected QT interval using Fridericia's formula (QTcF) prolongation at rest, where the mean QTc interval is > 480 msec based on triplicate measurements of electrocardiogram (ECG).
* Subject with stroke or other severe cerebrovascular diseases within 12 months before enrollment;
* Subject with interstitial lung disease or acute lung infection not yet recovered including but not limited to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection;
* Subject is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
adverse events | Through study completion, approximately 3 years
  Number of subjects participants with adverse events
Objective response rate (ORR) per RECIST v1.1 | Through study completion, approximately 3 years
  Defined as the proportion of patients with complete response (CR) or partial response (PR).

CONTACTS AND LOCATIONS:
Overall Officials: Zhengbo Song, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Cancer Hospital of the University of Chinese Academy of Sciences,, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No